CLINICAL TRIAL: NCT02957864
Title: Switching to Tenofovir Alafenamide Fumarate or Abacavir in Patients With Tenofovir Disoproxil Fumarate Associated eGFR Decline. A Randomized Trial.
Brief Title: Switching From Tenofovir Disoproxil Fumarate to Abacavir or Tenofovir Alafenamide
Acronym: BACTAF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Bart Rijnders, principle investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL55668.078.16
Record Dates: First submitted 2016-11-04; First posted 2016-11-08 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Renal Insufficiency,Chronic; Hiv; Therapeutic Agent Toxicity
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acquired Immunodeficiency Syndrome; Drug-Related Side Effects and Adverse Reactions | interventions — tenofovir alafenamide; emtricitabine tenofovir alafenamide; abacavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Switch to tenofovir alafenamide (Experimental): Switch from tenofovir disoproxil fumarate (TDF) to tenofovir alafenamide
  Interventions: Drug: tenofovir alafenamide
- Switch to abacavir (Active Comparator): Switch from tenofovir disoproxil fumarate (TDF) to abacavir
  Interventions: Drug: abacavir

INTERVENTIONS:
Drug: tenofovir alafenamide
  Other Names: Descovy; TAF
  Arms: Switch to tenofovir alafenamide
Drug: abacavir
  Other Names: ABC
  Arms: Switch to abacavir

SUMMARY:
Tenofovir disoproxil fumarate (TDF) is one of the most frequently used drugs to treat HIV. Long term use of TDF can induce renal toxicity. Tenofovir alafenamide (TAF) is a new pro-drug of Tenofovir which has not been associated with renal toxicity and may therefore be a good substitute for TDF in patients with TDF induced renal toxicity. Abacavir (ABC) is another drug that can be used for the treatment of HIV and is not associated with renal toxicity.

In this study the investigators will compare the effect on renal function of a switch from TDF to TAF with a switch from TDF to ABC in patients with TDF induced renal insufficiency.

DETAILED DESCRIPTION:
The majority of HIV-1 infected patients in resource rich countries receive the tenofovir prodrug tenofovir disoproxil fumarate (TDF) as part of their combination antiretroviral therapy (cART). Long-term exposure to TDF can be associated with an accelerated estimated glomerular filtration rate (eGFR) decline and proximal renal tubular dysfunction (PTD, see definition below). The current practice in patients in which TDF related renal toxicity becomes apparent is to substitute abacavir (ABC) for TDF. However, ABC is contraindicated in patients with HLAB57*01 and has been associated with an increased risk of cardiovascular disease in large HIV cohort studies, but not in randomized clinical trials. Recently, a new tenofovir prodrug, tenofovir alafenamide (TAF) was developed by Gilead Sciences and is available in a coformulation with emtricitabine (FTC). Due to the targeted delivery of tenofovir inside the CD4 positive cell by this prodrug, only 25 mg TAF is needed for the same antiviral effect observed in patients taking 250 mg of TDF and this lower TAF dose leads to 90% lower serum levels of tenofovir. In recently completed phase III studies in which patients with a normal kidney function where included, this lower tenofovir exposure in patients on TAF was shown to prevent off-target renal and bone toxicity in comparison with patients taking TDF. However, whether an already established TDF related renal toxicity in a HIV patient can be reversed after a switch to TAF, remains to be shown.

Objective:

To study the renal safety when HIV patients with TDF related renal toxicity switch to TAF compared to the current practice of switching to ABC.

Study design:

96 week open label multicenter randomized non-inferiority clinical trial.

Study population:

HIV-1 infected adults, suppressed HIV-RNA <50c/mL on a TDF containing antiretroviral regimen, with signs of TDF related renal toxicity as indicated by an accelerated eGFR decline.

Intervention:

Replace TDF with TAF (intervention arm) or ABC (control arm).

Main study parameters/endpoints:

Primary endpoint:

Recovery of renal dysfunction in the TAF arm versus the ABC arm at 48 weeks after the switch from TDF to TAF or ABC using the time to the first eGFR within 75% of the eGFR at the time of TDF initiation.

Secondary endpoints:

See below

ELIGIBILITY:
Inclusion Criteria:

HIV-positive documented by ELISA or Western Blot or plasma HIV-RNA > 1000 copies/mL.

18 years or older. Stable on TDF/FTC or TDF/3TC for ≥12 months (365 days) in combination with a third antiretroviral agent (NNRTI, INI, or PI) and with an unchanged third agent for at least 1 month.

HIV-1 RNA <50 copies/mL for ≥ 6 months. Patient is negative for the HLA B5701 allele.

Confirmed/probable TDF-related accelerated eGFR decline (one of the following):

1. Accelerated eGFR decline: mean of > 3 mL/min/year since start TDF after ≥5 years of TDF exposure.
2. Confirmed eGFR < 70 mL/min in patients with baseline eGFR > 90 mL/min at start of TDF.
3. eGFR decrease > 25% compared to baseline eGFR at TDF-initiation.

Absence of other causes of eGFR decline:

Diabetic patients with diabetic nephropathy (defined as an eGFR decline and uACR>30mg/mmol with uAPR >/=0.4, or biopsy proven).

Hypertensive patients (defined as the use of antihypertensives or untreated systolic (>=160mmHg) or diastolic (>=95mmHg) hypertension) in combination with hypertensive nephropathy (defined as eGFR decline with uACR>30mg/mmol with uAPR>/=0.4, or biopsy proven).

Nephrotic syndromes/nephrotic range proteinuria (uACR >300mg/mmol and uAPR ≥ 0.4, or total 24hrs proteinuria >3.5g/24hr, or biopsy proven) Nephrotic syndromes including rapid progressive glomerulonephritis and tubular interstitial nephritis (defined as active urine sediment with erythrocyturia and leucocyturia and proteinuria with eGFR decline, with or without the presence of systemic disease, or biopsy proven).

Obvious other renal toxic effects related to lifestyle or medication (e.g. creatin use) suspected by the investigators or biopsy proven.

Concomittantly used medication does not interfere with trial procedures (on investigators' discretion).

Exclusion Criteria:

Likely other cause (as defined above) of the accelerated GFR decline. HLA-B5701 positivity. Active hepatitis C or B. Documented intermediate or high level resistance to ABC. eGFR <30ml/min. Any other disease or medical condition that, in the opinion of the investigators, would interfere with the safety of the participant or the conduct of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-10; Primary Completion 2020-06 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Recovery of renal insufficiency | 48 weeks
  Recovery of renal dysfunction in the TAF arm versus the ABC arm at 48 weeks after the switch from TDF to TAF or ABC using the time to the first eGFR within 75% of the eGFR at the time of TDF initiation.

SECONDARY OUTCOMES:
Time to recovery of renal dysfunction | 96 weeks
  The between group differences (TAF vs ABC) with respect to the time to recovery of renal dysfunction (eGFR improvement to within 75% of eGFR at TDF initiation) at week 96, with adjustment for potentially important confounders.
Slope of eGFR-decline/increase | 96 weeks
  The mean eGFR at week 48 and 96 on ABC and TAF will be compared to week 0. The slopes of eGFR-decline/increase between week 0, week 48 and 96 will be compared between the ABC and TAF group.
Recovery of proteinuria | 96 weeks
  The median (IQR) of uPCR, uACR, uAPR, uB2MG/CR changes at week 48 and 96 compared to week 0 within the ABC and TAF group and difference in change between both groups.
Recovery of proximal tubular dysfunction | 96 weeks
  Changes in the number of patients with at least 2 markers of PTD from week 0 to week 48 within the ABC and TAF group and difference in change of PTD markers between both groups .
plasma HIV RNA <50c/ml | 96 weeks
  HIV-RNA suppression rate <50 ABC versus TAF at week 48 and 96.
Adverse events | 96 weeks
  Tolerability of TAF versus ABC, defined in terms of adverse events (%).
Framingham risk score | 96 weeks
  Change in framingham risk-score, blood pressure, lipids and inflammation parameters at week 0, 48 and 96 within the ABC and TAF group and comparison of between group differences of these parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Bart Rijnders, MD PhD, Study Director — Erasmus Medical Center
Locations (5):
- Netherlands (5):
  - Ziekenhuis Rijnstate, Arnhem, Gelderland
  - MC Slotervaart, Amsterdam
  - OLVG, Amsterdam
  - Erasmus MC, Rotterdam
  - Maasstad ziekenhuis, Rotterdam

IPD SHARING:
Plan to Share IPD: No